CLINICAL TRIAL: NCT03332615
Title: Motivational Interviewing to Address Reluctance and Ambivalence in Palliative Care
Brief Title: Motivational Interviewing in Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-1196
Record Dates: First submitted 2017-08-18; First posted 2017-11-06 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Motivational Interviewing
Keywords: Palliative Care
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinicians with MI coaching (Active Comparator): Clinicians in the intervention arm will be taught Motivational Interviewing via a coaching model in which a didactic session is followed by feedback through review of clinicians' audio-recorded encounters.
  Interventions: Behavioral: Motivational Interviewing
- Wait-list control (Placebo Comparator): After consent, clinicians in the wait-list control arm will complete a survey to self-assess their motivational interviewing skills and burnout.
  Interventions: Behavioral: Wait-list control

INTERVENTIONS:
Behavioral: Motivational Interviewing — Clinicians in the intervention arm will be taught Motivational Interviewing via a coaching model in which a didactic session is followed by feedback through review of clinicians' audio-recorded encounters.
  Arms: Clinicians with MI coaching
Behavioral: Wait-list control — After consent, clinicians in the wait-list control arm will complete a survey to self-assess their motivational interviewing skills and burnout.
  Arms: Wait-list control

SUMMARY:
Patients with advanced illness and their families confront a number of issues ranging from distressing symptoms to making complex decisions that affect quality of life and survival. Patients and family members struggle with these decisions even more when they feel ambivalence or reluctance. The investigator's overarching goal is to enhance provision of high quality, patient-centered care for patients with advance illness and their families and to reduce burnout among palliative care clinicians. The investigator will apply a well-established approach to achieving clinician/patient alignment in the primary care setting, Motivational Interviewing (MI) to a new population and setting, palliative care.

DETAILED DESCRIPTION:
The investigator will use a 2-arm randomized wait-list control design with up to 30 palliative care clinicians (15 in each arm). Clinicians in the intervention arm will be taught Motivational Interviewing (MI) via a coaching model in which a didactic session is followed by feedback through review of clinicians' audio-recorded encounters. Clinicians in both arms will audio record 4 encounters with patients with advanced illness and their family caregivers. The patients/caregivers will be provided with a 1-page information sheet about the study and will sign a HIPAA B form which will allow the study team to record a palliative care encounter and allow the research assistant to administer a short survey immediately within 1-2 days following a palliative care encounter to assess the effect of integrating MI techniques on perceived empathy and satisfaction with the encounter. The investigators will also assess clinician satisfaction with the encounter. Clinician burnout will be assessed at the time of study enrollment and following completion of all study encounter recordings. Clinicians randomized to the wait-list control arm will receive MI coaching only after they have recorded 4 study encounters. The wait-list control study design was selected to give all participating clinicians access to motivational interviewing coaching.

Intervention: The investigator is comparing standard palliative care communication skills enhanced by Motivational Interviewing coaching to standard palliative care. Given that palliative care is currently the gold standard for clinician communication in the setting of serious and advanced illness, if Motivational Interviewing coaching improves encounters for palliative care clinicians, it is even more likely to do so for other clinicians who care for people with advanced illness. The investigator has adopted a "coaching" model that includes both didactic and individual feedback. The coaching approach maps to Social Cognitive Theory in that its purpose is to build skills and improve self-efficacy or confidence to use the techniques. Participating palliative care clinicians randomized to the intervention arm will receive Motivational Interviewing coaching immediately. Those randomized to the wait-list control arm will receive Motivational Interviewing coaching after the study encounters and data collection have been completed. The intervention consists of several components: 1) 1-hour face-to-face (in person or via Skype) didactic session in which a Motivational Interviewing coach explains tenets of Motivational Interviewing and specifics, particularly addressing ambivalence and reluctance. This session will be recorded for future broader dissemination; 2) 1-hour individual session via Skype, including individualized goal-setting; 3) Clinician audio records 2 encounters, which are transcribed. The Motivational Interviewing coach then codes the encounters and meets with the clinician via Skype for 30 minutes to give feedback and coaching; 4) Clinician audio records 2 additional encounters and again receives individualized feedback and coaching. At the end of the interactive Motivational Interviewing didactic, each clinician who is randomized to the intervention arm will set an individual goal for which Motivational Interviewing technique he/she wants to try.

Each clinician will then audio record 2 palliative care encounters; audio recordings will be transcribed. The Motivational Interviewing coach will listen to the recordings and code the transcriptions paying attention to the clinician's stated goal. The coach will conduct 1:1 Skype calls to review audio-recorded encounters and provide individualized feedback and coaching. During the feedback sessions, the coach will provide positive feedback on the Motivational Interviewing techniques used, paying most attention to the technique the clinician set as his/her individual target technique. The coach will also offer feedback on parts of the encounter when Motivational Interviewing could have been applied. At the end of the session, the coach will ask the clinician to set another individual goal for which Motivational Interviewing technique they want to try and repeat the process of having them audio record 2 additional palliative care encounters and providing individualized feedback and coaching. After each clinician has finished the intervention, the investigators will obtain extensive process data from clinicians to learn what went well about the coaching and what can be improved to plan for future refinement and study. To plan for future scalability, the investigators will simultaneously be developing a coaching manual that will be used to train others to serve as Motivational Interviewing coaches.

Wait List Control: Clinicians who are randomized to the wait-list control arm will audio record 4 palliative care encounters, which will be transcribed, and have an individual coaching and feedback session in which the Motivational Interviewing coach will review their audio-recorded encounters following completion of study data collection.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians who are palliative care providers (physicians and Advanced Practice Providers).
* Patients/family caregivers must be 18 - 100 years of age.
* Patients must have an advanced illness and be receiving palliative care.
* Family caregivers must be caring for a patient who has an advanced illness who is receiving palliative care.

Exclusion Criteria:

* Patients/family caregivers who do not speak English or require interpreter services will be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Aim 1: feasibility and acceptability of learning Motivational Interviewing techniques by palliative care clinicians | Through study completion, an average of 1 year.
  To determine palliative care clinician-rated feasibility and acceptability of learning Motivational Interviewing techniques. Feasibility will be defined as the proportion of participating clinicians who successfully complete study participation (i.e. record 4 patient/caregiver encounters and provide post-test assessment).

SECONDARY OUTCOMES:
Aim 2: measure effects of the application of Motivational Interviewing techniques | Through study completion, an average of 1 year.
  To provide preliminary data on the effects of the application of Motivational Interviewing techniques on patient, caregiver and clinician perceptions of palliative care clinical encounters and on palliative care burnout. The investigator proposes to assess patient (or family caregiver)-reported Perceived Empathy and patient (or family caregiver) and clinician-reported Satisfaction with the palliative care encounter (within 2 days of the encounter). We will also assess clinician burnout prior to and following the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Jean S Kutner, MD, MSPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pollak KI, Gao X, Arnold RM, Arnett K, Felton S, Fairclough DL, Kutner JS. Feasibility of Using Communication Coaching to Teach Palliative Care Clinicians Motivational Interviewing. J Pain Symptom Manage. 2020 Apr;59(4):787-793. doi: 10.1016/j.jpainsymman.2019.11.010. Epub 2019 Nov 23. PMID 31765759